CLINICAL TRIAL: NCT04710511
Title: Association Between Child's Psychological Resilience and Practicing Oral Habits: Cross Sectional Study
Brief Title: Association Between Child's Psychological Resilience and Practicing Oral Habits
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mennat Allah Ashraf Abd Elsabour Abd Elkareem, Principle investigator, Cairo University
Other Study IDs: M111
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Oral Habits

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group: Medically free children aged from 5 years to 7 years and do not practice oral habits.
  Interventions: Other: Child and Youth Resilience Measure - Revised (CYRM-R)
- Oral habit practicing group: Medically free children aged from 5 years to 7 years and practicing oral habits.
  Interventions: Other: Child and Youth Resilience Measure - Revised (CYRM-R)

INTERVENTIONS:
Other: Child and Youth Resilience Measure - Revised (CYRM-R) — (CYRM-R): questionnaire , answered by the child (PMK): questionnaire, answered by the parent
  Other Names: Person Most Knowledgeable (PMK)

SUMMARY:
The aim of the present study is to determine the effect of psychological resilience on practicing oral habits among a group of 5- to 7-year-old children.

DETAILED DESCRIPTION:
Psychological pressure has been thought to be a predisposing factor that might result in deleterious oral habits practicing. Shahraki et al. stated that increased stress levels are associated with oral habits as thumb sucking and nail biting. Leme et al. concluded that children and adolescents with DOH presented more symptoms of depression than their counterparts. Moreover, they were more likely to report symptoms of anxiety.

Ability to cope (or resilience) includes a person's sense of agency and their ability to think and behave, to make positive decisions, and to apply skills and knowledge to life challenges. The term resilience has come to mean an individual's ability to overcome adversity and continue his or her normal development.

The association between psychological resilience and practicing oral habits in children remains unclear, this study aims to reveal that association, if present.

ELIGIBILITY:
Inclusion Criteria:

* Medically free children

Exclusion Criteria:

-

Ages: 5 Years to 7 Years | Sex: All
Age Groups: Child
Study Population: Medically free children aged from 5 years to 7 years
Sampling Method: Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Psychological resilience | Base line, subject will asked to fill the questionnaire for once
  Measured by: Child & Youth Resilience Measure - Revised It Consists of 17 questions answered by the child, choices optiones scored as (No = 1 , sometimes = 2, Yes = 3) The upper limit of the score is 51 and the lower limit is 17 the higher the score the higher the psychological resilience that the child has.

CONTACTS AND LOCATIONS:
Overall Officials: Mennat Allah A.Elkareem, B.D.S, Principal Investigator — Fuculty of Dentistry, Ahram Canadian University
Locations (1):
- This study is carried out online, through social media, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Subject age, gender, and his score in (CYRM-R) & (PMK) questionnaire.

REFERENCES:
- [Background] Leme M, Barbosa T, Castelo P, Gaviao MB. Associations between psychological factors and the presence of deleterious oral habits in children and adolescents. J Clin Pediatr Dent. 2014 Summer;38(4):313-7. doi: 10.17796/jcpd.38.4.c48238322205466w. PMID 25571681
- [Background] Measure, Y. R. (2011). Child and Youth Resilience Measure.
- [Background] Nicole, B., Velida, D.-S., & Michelle, R. (2018). Guidance on Measuring Children ' s Psychosocial Well - being. https://www.crs.org/sites/default/files/tools-research/meal4kids_well-being_guidance_aug_10_lo_res.pdf
- [Background] Resilience Research Centre. (2018). Child and Youth Resilience Measure (CYRM-R) & Adult Resilience Measure (ARM-R) Manual 2.2. CYRM and ARM User Manual. http://www.resilienceresearch.org/
- [Background] hahraki, N., Yassaei, S., & Moghadam, M. G. (2012). Abnormal oral habits: A review. Journal of Dentistry and Oral Hygiene, 4(May), 12-15. https://doi.org/10.5897/JDOH12.001